CLINICAL TRIAL: NCT00095056
Title: Sitagliptin Study in Patients With Type 2 Diabetes Mellitus and Chronic Renal Insufficiency
Brief Title: An Investigational Drug in Patients With Type 2 Diabetes Mellitus and Chronic Renal Insufficiency (0431-028)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-028; 2004_054
Record Dates: First submitted 2004-10-29; First posted 2004-11-01 (Estimated); Results first posted 2010-07-23 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2; Chronic Renal Insufficiency
Keywords: Type 2 Diabetes Mellitus and Chronic Renal Insufficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — Sitagliptin Phosphate; Glipizide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sitagliptin (Experimental): Participants in the Sitagliptin treatment sequence will receive sitagliptin in Phase A and placebo to glipizide in Phase B.
  Interventions: Drug: sitagliptin; Drug: glipizide; Drug: Placebo to glipizide
- Placebo (Placebo Comparator): Participants in the Placebo treatment sequence will receive placebo to sitagliptin in Phase A and glipizide in Phase B.
  Interventions: Drug: Placebo to Sitagliptin; Drug: glipizide

INTERVENTIONS:
Drug: sitagliptin — One (participants with visit 1 estimated creatinine clearance <30 mL/min or undergo regular dialysis) or Two (participants with visit 1 creatinine clearance of =30 to <50 mL/min; not on dialysis) tablets of 25 mg Sitagliptin daily.
  Other Names: MK0431
  Arms: Sitagliptin
Drug: Placebo to Sitagliptin — One (participants with visit 1 estimated creatinine clearance <30 mL/min or undergo regular dialysis) or Two (participants with visit 1 creatinine clearance of =30 to <50 mL/min and not on dialysis) tablets of placebo to sitagliptin 25 mg daily.
  Arms: Placebo
Drug: glipizide — One 5 mg glipizide tablet per day. The dose of glipizide administered per day may be increased after 2 weeks and at 2-week intervals thereafter up to 20 mg based upon fingerstick glucose determinations.
Drug: Placebo to glipizide — One placebo to glipizide 5 mg tablet per day. The dose of placebo to glipizide administered per day may be increased after 2 weeks and at 2-week intervals thereafter up to 20 mg based upon fingerstick glucose determinations.
  Arms: Sitagliptin

SUMMARY:
The purpose of this study is to determine the safety and tolerability of an investigational drug in patients with Type 2 Diabetes Mellitus (a specific type of diabetes) and Chronic Renal Insufficiency (inadequate kidney function).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age diagnosed with type 2 diabetes mellitus (T2DM) (a specific type of diabetes).
* Patient has renal (kidney) insufficiency (inadequate kidney function)

Exclusion Criteria:

* Patient has had heart problems (such as a heart attack or chest pain) or stroke within the past 6 months or any condition or therapy which, in the opinion of the investigator, may not be in the patient's best interest to participate.
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2004-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Chan JC, Scott R, Arjona Ferreira JC, Sheng D, Gonzalez E, Davies MJ, Stein PP, Kaufman KD, Amatruda JM, Williams-Herman D. Safety and efficacy of sitagliptin in patients with type 2 diabetes and chronic renal insufficiency. Diabetes Obes Metab. 2008 Jul;10(7):545-55. doi: 10.1111/j.1463-1326.2008.00914.x. Epub 2008 Jun 1. PMID 18518892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 14-Dec-04
  Last Patient Last Visit: 27-Jul-06
  75 study centers worldwide
Pre-assignment Details: Patients ≥18 years of age with chronic renal insufficiency and type 2 diabetes mellitus who had an A1C of 6.5-10% (not on baseline insulin therapy) or 7.5-10% (on baseline insulin therapy) after an antihyperglycemic agent (AHA) wash-off period of up to 12 weeks, were eligible to enter the 54-week
  study.
Groups:
- Sitagliptin: The Sitagliptin group includes data from patients randomized to receive treatment with either one (1) 25 mg oral tablet of sitagliptin once daily (blinded) [patients with Creatinine Clearance (CrCl) <30 mL/min or dialysis] or two (2) 25 mg oral tablets of sitagliptin once daily (blinded) [patients with CrCl 30 to <50mL/min] alone or in combination with baseline insulin therapy. During Phase B, patients in the Sitagliptin group (with the exception of patients on baseline insulin therapy and patients who received glycemic rescue medication in Phase A) were given glipizide placebo (blinded). During Phase B, patients on baseline insulin could have their insulin uptitrated, and patients who received glycemic rescue medication in Phase A continued on open-label rescue medication.
- Placebo: The Placebo group includes data from patients randomized to receive treatment with either one (1) tablet of placebo matching sitagliptin 25 mg (blinded) [patients with CrCl <30 mL/min or dialysis] or two (2) tablets of placebo matching sitagliptin 25 mg (blinded) [patients with CrCl 30 to <50mL/min] alone or in combination with baseline insulin therapy. During Phase B, patients in the Placebo group (with the exception of patients on baseline insulin therapy and patients who received glycemic rescue medication in Phase A) were given glipizide (blinded). During Phase B, patients on baseline insulin could have their insulin uptitrated, and patients who received glycemic rescue medication in Phase A continued on open-label rescue medication.
Period: Phase A (Weeks 0-12)
Arm/Group | Sitagliptin | Placebo
Started | 65 | 26
Completed | 58 | 25
Not Completed | 7 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Death | 1 | 0
Not completed — Protocol specific criteria | 2 | 0
Period: Phase B (Weeks 12-54)
Arm/Group | Sitagliptin | Placebo
Started | 56 (2 randomized patients completed Period 1 but did not enter Period 2.) | 25
Completed | 46 | 20
Not Completed | 10 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Patient Moved | 1 | 0
Not completed — Death | 3 | 1
Not completed — Protocol specific criteria | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 65 | 26 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (9.8) | 65.3 (9.7) | 67.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 10 | 44
  Male | 31 | 16 | 47
Race/Ethnicity, Customized [Number; unit: participants]
  White | 22 | 8 | 30
  Black | 4 | 1 | 5
  Hispanic | 17 | 9 | 26
  Asian | 20 | 7 | 27
  Other | 2 | 1 | 3
HbA1c (Hemoglobin A1c) [Mean (Standard Deviation); unit: Percent] | 7.6 (0.9) | 7.8 (0.9) | 7.7 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Sitagliptin After 12 Weeks of Treatment
Description: Safety and tolerability were measured in terms of the number of patients with clinical adverse experiences (CAEs), serious CAEs, drug-related CAEs, laboratory adverse experiences (LAEs), serious LAEs, and drug-related LAEs. Drug-relationship was assessed by the study investigator according to his/her best clinical judgment.
Time Frame: Week 0 through Week 12
Population: All patients who took study medication were included in the analysis. Events that occurred after initiation of glycemic rescue therapy were excluded from the analysis of CAEs, drug-related CAEs, LAEs, & drug-related LAEs. Events that occurred after initiation of glycemic rescue therapy were included in the analysis of serious CAEs and serious LAEs.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 65 | 26
Participants
  With CAEs | 41 | 16
  With drug-related CAEs | 8 | 1
  With serious CAEs | 9 | 1
  With LAEs | 9 | 5
  With drug-related LAEs | 1 | 0
  With serious LAEs | 0 | 0

2. Secondary Outcome: Safety and Tolerability of Sitagliptin Over 54 Weeks
Description: as for outcome 1
Time Frame: Week 0 through Week 54
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 65 | 26
Participants
  With CAEs | 50 | 22
  With drug-related CAEs | 8 | 5
  With serious CAEs | 20 | 10
  With LAEs | 15 | 8
  With drug-related LAEs | 2 | 0
  With serious LAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 0 through Week 54
Description: Patients received rescue medication if they met specific glycemic goals. This summary of SAEs includes events that occurred either before or after receiving rescue medication. This summary of Other AEs includes only those AEs that occurred prior to a patient receiving rescue medication.
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 20/65 | 10/26
Other Adverse Events (participants affected / at risk) | 29/65 | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=65) | Placebo (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0
Cardiac Failure (Cardiac disorders) | 2 | 0
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Retinopathy (Eye disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Sudden Death (General disorders) | 1 | 0
Arteriovenous Graft Site Infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 2 | 0
Septic Shock (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 1
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Polytraumatism (Injury, poisoning and procedural complications) | 0 | 1
Diabetic Foot (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 1 | 0
Thalamic Infarction (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 1
Renal Failure Chronic (Renal and urinary disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Hypertensive Crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=65) | Placebo (N=26)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 2
Oedema Peripheral (General disorders) | 2 | 2
Catheter Site Infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 4 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 5
Urinary Tract Infection (Infections and infestations) | 5 | 3
Blood Creatinine Increased (Investigations) | 1 | 2
Blood Glucose Increased (Investigations) | 3 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.